CLINICAL TRIAL: NCT02196818
Title: A Multi-centre, Prospective Post Marketing Surveillance Study to Assess Mid-term Performance of the Mpact Cup in Subjects Requiring Primary Total Hip Arthroplasty
Brief Title: A Multi-centre, Prospective Surveillance to Assess Mid-term Performance of the Mpact Cup
Status: Terminated | Type: Observational
Why Stopped: Study was closed mainly because the surgeons participating no longer had the infrastructure to support the research and weren't following their subjects
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P01.014.08/00
Record Dates: First submitted 2014-07-07; First posted 2014-07-22 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Osteoarthritis; Arthritis; Avascular Necrosis; Fracture of the Femoral Neck or Head; Congenital Hip Dysplasia
MeSH Terms: conditions — Osteoarthritis; Arthritis; Osteonecrosis; Hip Dislocation, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Mpact Acetabular Shell: Monitor the performance of the Mpact cup in the treatment of patients with hip joint disease requiring a total hip replacement.
  Interventions: Device: Mpact Acetabular Shell

INTERVENTIONS:
Device: Mpact Acetabular Shell — Total Hip Replacement

SUMMARY:
This is a multi-centre, prospective post marketing surveillance study to assess mid-term performance of the Mpact cup in subjects requiring primary total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are willing and able to provide written informed consent for participation in the study. Written informed consent must be obtained prior to the patient's surgery.
* Those presenting with disease that meets the indications for use for Medacta USA implants defined by this study (on-label use).
* Patients must be willing to comply with the pre and post-operative evaluation schedule.

Exclusion Criteria:

* Those with one or more medical conditions identified as a contraindication defined by the labeling on any Medacta implants used in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary total hip arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
The Kaplan-Meier analysis as a measure of implant performance. | 5 years

SECONDARY OUTCOMES:
The Harris Hip Score. | pre-op, 3/6 months, 1,2 and 5 years
Radiological analysis as a meausure of safety. | 3/6 months, 1,2 and 5 years

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Vail Orthopedics, P.C., Denver, Colorado
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Illinois Bone & Joint Institute, LLC, Libertyville, Illinois
  - Jordan Valley Medical Center, West Jordan, Utah